CLINICAL TRIAL: NCT01938248
Title: Apixaban for the Reduction of Thrombo-Embolism in Patients With Device-Detected Sub-Clinical Atrial Fibrillation
Acronym: ARTESiA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry); Pfizer (Industry); Medtronic (Industry); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Jeff Healey, Principal Investigator, Population Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ARTESiA; 2014-001397-33 (EudraCT Number)
Record Dates: First submitted 2013-09-04; First posted 2013-09-10 (Estimated); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Atrial Fibrillation; Stroke
Keywords: Pacemaker, Artificial; Defibrillators, Implantable; Atrial Fibrillation; Stroke Risk
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — apixaban; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Aspirin 81 mg once daily
  Interventions: Drug: aspirin
- Intervention (Experimental): Apixaban, 5 mg twice daily (or 2.5 mg twice daily if 2 or more of: age > 80, weight ≤ 60 kg or serum creatinine ≥ 133 mmol/L)
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban — apixaban at a dose of 5 mg twice daily (2.5 mg twice daily if 2 or more of: age > 80, weight ≤ 60 kg or serum creatinine ≥ 133 mmol/L)
  Other Names: Eliquis
  Arms: Intervention
Drug: aspirin — aspirin 81 mg once daily
  Other Names: ASA; acetylsalicylic acid
  Arms: Control

SUMMARY:
This study aims to determine if treatment with apixaban, compared with aspirin, will reduce the risk of ischemic stroke and systemic embolism in patients with device-detected sub-clinical atrial fibrillation and additional risk factors for stroke.

DETAILED DESCRIPTION:
Device-detected sub-clinical atrial fibrillation (SCAF) is a new disorder that has been recognized since the availability of implantable devices capable of long term continuous heart rhythm monitoring. It is characterized by one or more runs of rapid atrial arrhythmia detected by the device without symptoms and without any clinical atrial fibrillation (AF) detected by the usual methods, (i.e. electrocardiogram, Holter monitor, etc.). In the ASSERT trial, SCAF was detected by a pacemaker or implantable cardioverter defibrillator (ICD) in nearly 40% of patients during 2 and a half years of follow up. The presence of SCAF increased stroke risk by 2.5-fold (1). The risk of stroke or systemic embolism among patients with SCAF and a CHADS2 score ≥ 4 was 2.75% per year. Oral anticoagulation is effective and safe for stroke prevention in patients with clinical atrial fibrillation, but it is unknown if the same risk benefit ratio exists for anticoagulation therapy in patients with SCAF (2;3). SCAF differs from clinical AF in being of shorter duration, being asymptomatic, and often have a more regular rhythm in the right atrium where it is typically detected. Data ASSERT suggest that the increase in stroke risk with SCAF may be less than the increase with clinical AF. Therefore opinion leaders have written that the role of oral anticoagulation for the treatment of SCAF is uncertain and that randomized trials of anticoagulation are needed (4;5). Recent surveys of pacemaker clinic practice indicate that only 25% of patients with SCAF are treated with oral anticoagulation (6;7). Thus there is clinical equipoise for a trial of oral anticoagulation compared to aspirin in higher risk patients with SCAF.

Apixaban is a Factor Xa inhibitor that is an effective and safe anticoagulant. It has been shown to have an excellent risk benefit profile for stroke prevention in clinical AF (14, 15). It is highly suitable to test if oral anticoagulation therapy will reduce the risk of stroke or systemic embolism in SCAF.

Patients will be randomized double-blind to receive apixaban or aspirin. Apixaban dose will be 5 mg twice daily (2.5 mg twice daily if 2 or more of: age > 80, weight ≤ 60 kg or serum creatinine ≥ 133 mmol/L). Those assigned to aspirin will receive a dose of 81 mg daily. The study will be event driven and will continue until 248 patients have experienced a primary outcome event.

ELIGIBILITY:
Inclusion Criteria:

1. Permanent pacemaker or defibrillator (with or without resynchronization) or insertable cardiac monitor capable of detecting SCAF
2. At least one episode of SCAF ≥ 6 minutes in duration but no single episode > 24 hours in duration at any time prior to enrollment. Any atrial high rate episode with average > 175 beats/min will be considered as SCAF. No distinction will be made between atrial fibrillation and atrial flutter. SCAF requires electrogram confirmation (at least one episode) unless ≥ 6 hours in duration.
3. Age ≥ 55 years
4. Risk Factor(s) for Stroke:

Previous stroke, TIA or systemic arterial embolism OR Age at least 75 OR Age 65-74 with at least 2 other risk factors OR Age 55-64 with at least 3 other risk factors

Other risk factors are:

* hypertension
* CHF
* diabetes
* vascular disease (i.e. CAD, PAD or Aortic Plaque)
* female

Exclusion Criteria:

1. Clinical atrial fibrillation documented by surface ECG (12 lead ECG, Telemetry, Holter) lasting ≥ 6 minutes, with or without clinical symptoms
2. Mechanical valve prosthesis, deep vein thrombosis, recent pulmonary embolism or other condition requiring treatment with an anticoagulant
3. Contra-indication to apixaban or aspirin:

   1. Allergy to aspirin or apixaban
   2. Severe renal insufficiency (creatinine clearance must be calculated in all patients; any patient with either a serum creatinine > 2.5 mg/dL [221 µmol/L] or a calculated creatinine clearance < 25 ml/min is excluded)
   3. Serious bleeding in the last 6 months or at high risk of bleeding (this includes, but is not limited to: prior intracranial hemorrhage, active peptic ulcer disease, platelet count < 50,000/mm3 or hemoglobin < 10 g/dL, recent stroke within past 10 days, documented hemorrhagic tendencies or blood dyscrasias)
   4. Moderate to severe hepatic impairment
   5. Ongoing need for combination therapy with aspirin and clopidogrel (or other combination of two platelet inhibitors)
   6. Meets criteria for requiring lower dose of apixaban AND also has ongoing need for strong inhibitors of CYP 3A4 or P-glycoprotein (e.g., ketoconazole, itraconazole, ritonavir or clarithromycin)
   7. Ongoing need for strong dual inducers of CYP 3A4 or P-glycoprotein (e.g., rifampin, carbamazepine, phenytoin, St. John's wort)
4. Received an investigational drug in the past 30 days
5. Participants considered by the investigator to be unsuitable for the study for any of the following reasons:

   1. Not agreeable for treatment with either aspirin or apixaban or anticipated to have poor compliance on study drug treatment
   2. Unwilling to attend study follow-up visits
   3. Life expectancy less than the expected duration of the trial2 years due to concomitant disease
6. Women who are pregnant, breast-feeding or of child-bearing potential without an acceptable form of contraception in place (sterilization, hormonal contraceptives, intrauterine device, barrier methods or abstinence)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4012 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-11-03 (Actual)

PRIMARY OUTCOMES:
Composite of ischemic stroke and systemic embolism | event driven, duration of follow-up - mean follow-up time anticipated: 3 years
  Definition of stroke:
  1. Rapid onset* of a focal/global neurological deficit
  2. Duration of a focal/global neurological deficit ≥ 24 hours OR the neurological deficit results in death OR the neurological deficit is supported by clear evidence of cerebral infarction on diffusion-weighted MRI imaging.
  3. No other readily identifiable non-stroke cause for the clinical presentation
  4. Confirmation of the diagnosis by specialist evaluation or brain imaging procedure
  Definition of Systemic Embolism:
  Clinical signs and symptoms consistent with embolic arterial occlusion plus at least one of the following objective findings of arterial embolism:
  * Surgical report indicating evidence of arterial embolism
  * Pathological specimens related to embolism removal
  * Imaging evidence consistent with arterial embolism
  * Autopsy reports
Major Bleed | duration of follow-up
  The main safety outcome will be the occurrence of clinically overt major bleeding as defined by the ISTH criteria:
  1. Fatal bleeding, and/or
  2. Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome, and/or
  3. Bleeding causing a fall in hemoglobin level of 2 g/dL or more, or leading to transfusion of two or more units of whole blood or red cells.

SECONDARY OUTCOMES:
Ischemic Stroke | Duration of Follow-up
Myocardial Infarction | Duration of follow-up
  MI definition:
  1. Typical rise and gradual fall (troponin) or more rapid rise and fall (CKMB) of biochemical markers of myocardial necrosis with at least one of: a) ischemic symptoms; b) development of pathological Q-waves on the ECG; c) ECG changes indicative of ischemia; d) Coronary artery intervention
     OR
  2. Pathological findings of an acute myocardial infarction
Cardiovascular Death | Duration of follow-up
All-cause Death | Duration of follow-up
Composite of stroke, MI, SE and death | Duration of follow-up
  Composite of stroke, myocardial infarction, systemic embolism and all-cause death
Composite of stroke, MI, SE, death and major bleeding | Duration of follow-up
  Composite of stroke, myocardial infarction, systemic embolism, all-cause death and major bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Healey, M.D., Principal Investigator — Population Health Research Institute; Stuart Connolly, M.D., Study Chair — Population Health Research Institute; Marco Alings, M.D., Principal Investigator — Working Group Cardiovascular Research Netherlands; Renato Lopes, M.D., Principal Investigator — Duke Clinical Research Institute
Locations (130):
- United States (23):
  - Cardiovascular Associates of Mesa, PC, Mesa, Arizona
  - St. Vincent Heart Clinic, Little Rock, Arkansas
  - Cardiovascular Associates of Marin and San Francisco Medical, Larkspur, California
  - Aurora Denver Cardiology Associates, Aurora, Colorado
  - Naples Interventional Cardiac Electrophysiology, Naples, Florida
  - Langhorne Cardiology Consultants, Inc., Pensacola, Florida
  - One Health Cardiology, Owensboro Health, Inc., Owensboro, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Michigan Heart, Ypsilanti, Michigan
  - University of Missouri Health System, Columbia, Missouri
  - St. Louis Heart and Vascular, St Louis, Missouri
  - Glacier View Cardiology, Kalispell, Montana
  - The Cooper Health System, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - St. Peter's Health Partners Medical Association, PC, Albany, New York
  - Carolinas Healthcare System, Charlotte, North Carolina
  - WakeMed, Raleigh, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Pennsylvania State University, Hershey, Pennsylvania
  - Research Institute of LG Health / Penn Medicine, Lancaster, Pennsylvania
  - Virginia Heart, Falls Church, Virginia
- Belgium (10):
  - Onze Lieve Vrouw Ziekenhuis, Aalst
  - Vivalia CSL St. Joseph, Arlon
  - Clinique Saint Jean-Brussels, Brussels
  - Grand Hopital de Charleroi, Gilly
  - AZ Groeninge, Kortrijk
  - University Hospitals Leuven, Leuven
  - CHC Saint Joseph, Liège
  - CHR de la Citadelle, Liège
  - AZ Delta, Roeselare
  - CHU Dinant-Godinne, Yvoir
- Canada (24):
  - University of Calgary Foothills Hospital, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Grey Nuns Hospital, Edmonton, Alberta
  - Heart Rhythm Research Office - St. Paul's Hospital, Vancouver, British Columbia
  - Victoria Cardiac Arrhythmia Trials, Inc., Victoria, British Columbia
  - St. Boniface Hospital, Winnepeg, Manitoba
  - Capital District Health Authority, Halifax, Nova Scotia
  - Health Sciences North, Greater Sudbury, Ontario
  - Hamilton General Hospital, Hamilton, Ontario
  - St. Mary's General Hospital, Kitchener, Ontario
  - London Health Sciences Centre, London, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Oakville Cardiologists, Oakville, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Sunnybrook Hospital, Toronto, Ontario
  - Institute Universitaire de Cardiologie and de Pneumonologie, Laval, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - CHUM - Hotel Dieu, Montreal, Quebec
  - Hopital Sacre-Coeur de Montreal, Montreal, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - CHUS - Sherbrooke, Sherbrooke, Quebec
  - Ciusss McQ, Trois-Rivières, Quebec
- IKEM Institute for Clinical and Experimental Medicine, Prague, Czechia
- Denmark (7):
  - Hilleroed Hospital, Hilleroed, North Zealand
  - Sygehus Sonderjylland, Aabenraa
  - Aalborg University Hospital, Dept of Cardiology, Aalborg
  - Aarhus Unniversity Hospital, Skejby, Aarhus
  - Gentofte Hospital, Hellerup
  - Odense University Hospital, Odense
  - Hjertemedicinsk Forskning, RH Viborg, HEM, Viborg
- Germany (8):
  - Johann Wolfgang Goethe University Hospital Frankfurt, Frankfurt am Main, Hesse
  - Katholisches Klinikum Mainz, Mainz, Rhineland-Palatinate
  - Universitatsklinikum des Saarlandes, Homburg/Saar, Saarland
  - MVZ am Kuchwald GmbH, Chemnitz, Saxony
  - Zentrum fur klinische Prufungen in der Facharztzentrum Dresd, Dresden, Saxony
  - University Medicine Gottingen, Göttingen
  - Asklepios Klinik Barmbek, Hamburg
  - Universitaetsklinikum Tuebingen, Kardiologie, Tübingen
- Hungary (3):
  - Allami Szivkorhaz Balatonfured, Balatonfüred, Veszprém megye
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Semmelweis University, Budapest
- Italy (10):
  - Ospedale Sant'Anna, San Fermo Della Batt, Como
  - Cardiologia-A.O. Desio e Vimercate - Presisio di Vimercat, Vimercate, Monza Brianza MB
  - Hospital Santa Maria Della Pieta, Nola, Napoli
  - AOU Ospedali Riuniti, Ancona
  - Ospedale Maggiore, Cardiologia Dept., Bologna
  - S.Orsola-Malpighi, Bologna
  - Bolzano Regional Hospital, Dept of Cardiology, Bolzano
  - Azienda Ospedaliero-Univeritaria Di Modena-Policlinico, Modena
  - Ospedale G.B. Grassi, Rome
  - University and Hospital of Trieste, Trieste
- Netherlands (15):
  - Gelre Ziekenhuis, Zutphen, Gelderland
  - Atrium Orbis Heerlen, Heerlen, Limburg
  - Amphia Hospital Breda, Breda, North Brabant
  - Ziekenhuis Tjongerschans, Heerenveen, Provincie Friesland
  - Ikazia Ziekenhuis, Rotterdam, South Holland
  - BovenIJ Ziekenhuis, Amsterdam
  - Hospital Rijnstate, Arnhem
  - Deventer Hospital, Cardiology Research, Deventer
  - Hospital Gelderse Vallei, Ede
  - Treant Hospital Department Cardiology, Emmen
  - Admiraal de Ruyter Ziekenhuis, Goes
  - Treant Hospital - Bethseda, Hoogeveen, Hoogeveen
  - Bravis Ziekenhuis, locatie Roosendaal, Roosendaal
  - (ETZ) Elisabeth Tweesteden Hospital, Tilburg
  - Máxima Medisch Centrum, Veldhoven
- Norway (2):
  - Barum Hospital, Vestre Viken, Drammen, Buskerud
  - Oslo University Hospital - Ulleval, Oslo
- Spain (13):
  - Hospital Clinico Santiago de Compostela, Santiago de Composte, A Coruna
  - Rafael Mendez Universitary Hospital, Lorca, Murcia
  - Complexo Hospitalario Universitario A Coruna, A Coruña
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Del Mar, Barcelona
  - Hospital Juan Ramon Jimenez, Huelva
  - Hospital Clinico San Carlos, Unidad De Arritmias, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Puerta de Hierro Majadahonda, Majadahonda
  - Agencia Sanitaria Costa del Sol- Hospital Costa del Sol, Marbella
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
- Switzerland (5):
  - University Hospital Basel, Basel, Canton of Basel-City
  - Kantonsspital St Gallen, Sankt Gallen, Canton of St. Gallen
  - CHUV, Lausanne, Canton of Vaud
  - Hopital Fribourgeois, site de Fribourg, Fribourg
  - University Hospital of Geneva, Geneva
- United Kingdom (9):
  - Dorset County Hospital NHS Foundation Trust, Dorchester, Dorset
  - Hampshire Hospitals (NHS Foundation Trust), Basingstoke, Hampshire
  - Portsmouth Hospitals NHS Trust, Portsmouth, Hampshire
  - Royal Alexandra Hospital, Paisley, Renfrewshire
  - Shrewsbury & Telford Hospital NHS, Shropshire, West Midlands
  - Blackpool Teaching Hospitals NHS Foundation Trust, Blackpool
  - Queen Elizabeth University Hospital, Glasgow
  - Liverpool Heart and Chest Hospital, Liverpool
  - Freeman Hospital, Newcastle upon Tyne

REFERENCES:
- [Derived] Siegal DM, Sticherling C, Healey JS, McIntyre WF, Christensen LS, Parkash R, Vanassche T, Conen D, Gold M, Granger CB, Nielsen JC, Carrier M, Wojdyla DM, Erath JW, Rivard L, Kutyifa V, Wright DJ, Lopes RD. Major Bleeding With Apixaban vs Aspirin: A Subanalysis of the ARTESiA Randomized Clinical Trial. JAMA Cardiol. 2025 Dec 1;10(12):1305-1314. doi: 10.1001/jamacardio.2025.4151. PMID 41222953
- [Derived] Shoamanesh A, Field TS, Coutts SB, Sharma M, Gladstone D, Hart RG, Boriani G, Wright DJ, Sticherling C, Birnie DH, Gold MR, Erath JW, Kutyifa V, Mian R, Benz AP, Granger CB, McIntyre WF, Connolly SJ, Nielsen JC, Alings M, Rivard L, Lopes RD, Healey JS; ARTESiA study investigators. Apixaban versus aspirin for stroke prevention in people with subclinical atrial fibrillation and a history of stroke or transient ischaemic attack: subgroup analysis of the ARTESiA randomised controlled trial. Lancet Neurol. 2025 Feb;24(2):140-151. doi: 10.1016/S1474-4422(24)00475-7. PMID 39862882
- [Derived] McIntyre WF, Benz AP, Healey JS, Connolly SJ, Yang M, Lee SF, Field TS, Alings M, Benezet-Mazuecos J, Boriani G, Nielsen JC, Gold MR, Pergolini F, Glotzer TV, Granger CB, Lopes RD. Risk of Stroke or Systemic Embolism According to Baseline Frequency and Duration of Subclinical Atrial Fibrillation: Insights From the ARTESiA Trial. Circulation. 2024 Nov 26;150(22):1747-1755. doi: 10.1161/CIRCULATIONAHA.124.069903. Epub 2024 Sep 4. PMID 39229707
- [Derived] Lopes RD, Granger CB, Wojdyla DM, McIntyre WF, Alings M, Mani T, Ramasundarahettige C, Rivard L, Atar D, Birnie DH, Boriani G, Amit G, Leong-Sit P, Rinne C, Duray GZ, Gold MR, Hohnloser SH, Kutyifa V, Benezet-Mazuecos J, Cosedis Nielsen J, Sticherling C, Benz AP, Linde C, Kautzner J, Mabo P, Mairesse GH, Connolly SJ, Healey JS. Apixaban vs Aspirin According to CHA2DS2-VASc Score in Subclinical Atrial Fibrillation: Insights From ARTESiA. J Am Coll Cardiol. 2024 Jul 23;84(4):354-364. doi: 10.1016/j.jacc.2024.05.002. Epub 2024 May 19. PMID 39019530
- [Derived] Healey JS, Lopes RD, Granger CB, Alings M, Rivard L, McIntyre WF, Atar D, Birnie DH, Boriani G, Camm AJ, Conen D, Erath JW, Gold MR, Hohnloser SH, Ip J, Kautzner J, Kutyifa V, Linde C, Mabo P, Mairesse G, Benezet Mazuecos J, Cosedis Nielsen J, Philippon F, Proietti M, Sticherling C, Wong JA, Wright DJ, Zarraga IG, Coutts SB, Kaplan A, Pombo M, Ayala-Paredes F, Xu L, Simek K, Nevills S, Mian R, Connolly SJ; ARTESIA Investigators. Apixaban for Stroke Prevention in Subclinical Atrial Fibrillation. N Engl J Med. 2024 Jan 11;390(2):107-117. doi: 10.1056/NEJMoa2310234. Epub 2023 Nov 12. PMID 37952132